CLINICAL TRIAL: NCT07277036
Title: The Effect of Video-Assisted Education on Postoperative Outcomes After Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Video-Assisted Education After Laparoscopic Cholecystectomy
Acronym: VAE-LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Tinaztepe University (Other)
Responsible Party: Principal Investigator, Berna Dizer, Assistant professor, Izmir Tinaztepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İzmirTınaztepeÜ-B.Dizer-002
Record Dates: First submitted 2025-11-19; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Laparoscopic Cholecystectomy; Patient Education
Keywords: Video-assisted education; patient education; defecation; self-care; postoperative recovery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-Assisted Education (Experimental): Single-session video-assisted patient education in addition to routine postoperative instructions
  Interventions: Behavioral: Video-Assisted Patient Education
- Usual Care (No Intervention): Routine postoperative discharge education without the video component.

INTERVENTIONS:
Behavioral: Video-Assisted Patient Education — Single-session video-assisted patient education delivered before hospital discharge after laparoscopic cholecystectomy. A standardized 10-15-minute video (shown on a tablet/TV by a nurse) covers postoperative care: pain control/analgesic use, early mobilization, wound care, diet/fluids, warning signs, and follow-up. Participants also receive routine discharge instructions; the video is an adjunct unique to this arm and is not provided to the control group.
  Arms: Video-Assisted Education

SUMMARY:
Brief Summary:

This randomized controlled trial aims to evaluate the effects of video-assisted preoperative education on postoperative physiological parameters and recovery outcomes in patients undergoing laparoscopic cholecystectomy. The study compares a video-based education program with brochure-based education covering pain and nausea-vomiting management, nutrition, early mobilization, fluid intake, wound care, bathing, and follow-up instructions in adults scheduled for elective laparoscopic cholecystectomy in a public state hospital in Türkiye.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is a widely used minimally invasive surgical method to treat gallstones. Effective preoperative education is critical to enhance postoperative recovery and reduce complications. This randomized controlled trial was conducted between October 1, 2023, and January 17, 2024, in the General Surgery Department of a public state hospital in Türkiye. The primary aim of the study is to determine the effects of video-assisted education on postoperative physiological parameters and recovery outcomes of patients undergoing laparoscopic cholecystectomy. A total of 92 adult patients scheduled for elective laparoscopic cholecystectomy are randomly assigned to an intervention group (n = 46) and a control group (n = 46) using a randomized allocation procedure. The intervention group receives structured video-assisted education, whereas the control group receives the same educational content through a printed brochure. The educational content includes information on postoperative pain and nausea-vomiting management, nutrition, early mobilization, adequate fluid intake, wound care, bathing, and follow-up instructions. Education is delivered preoperatively by a trained nurse.

Data are collected using a sociodemographic data form, the Visual Analog Scale (VAS) for pain, a pre-/postoperative patient assessment form, and a dietary habits questionnaire. Physiological parameters (vital signs, SpO₂, blood glucose), functional recovery indicators (defecation, mobilization, bathing), and selected self-care behaviors are assessed at predefined time points (preoperative baseline, discharge day, and postoperative follow-up day).

The primary outcomes are postoperative bowel recovery (e.g., presence and timing of defecation) and selected self-care-related recovery indicators (e.g., bathing status, need for family assistance). Secondary outcomes include postoperative nausea-vomiting, pain intensity, vital signs, and dietary habits. The study is designed to inform nursing practice regarding the use of video-assisted education compared with brochure-based education in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) undergoing elective laparoscopic cholecystectomy at the study hospital.
* Able to provide written informed consent and to receive/understand the education materials.
* Willing to complete postoperative assessments at discharge and on postoperative day 5-7

Exclusion Criteria:

* Impaired consciousness, speech difficulties, hearing impairment, or diagnosed psychiatric conditions that would preclude receiving the educational intervention or valid assessment.

(Operational exclusions after enrollment): cancellation of surgery, refusal to continue participation, or incomplete data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 92 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
Defecation Occurrence | Postoperative day 5-7 (follow-up)
  Proportion of participants who report at least one bowel movement by the follow-up day, recorded via the standardized patient assessment form. Higher proportions indicate faster gastrointestinal recovery. Groups compared: Video-Assisted Education vs. Usual Care

SECONDARY OUTCOMES:
Postoperative Nausea and Vomiting (Yes/No) | At hospital discharge (postoperative day 0-1).
  Any nausea or ≥1 vomiting episode on the day of discharge; proportions compared between groups.

OTHER OUTCOMES:
Bathing With Family Assistance (Yes/No) | Postoperative day 5-7 (follow-up)
  Need for family assistance during bathing at follow-up; proportions compared between groups.
Pain Intensity | At hospital discharge (postoperative day 0-1).
  Mean VAS pain score (0=no pain, 10=worst pain); higher scores indicate worse pain

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Tinaztepe University, Izmir, Buca, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The informed consent/IRB approval did not include permission for public deposition of individual participant-level data. In accordance with local privacy regulations (e.g., Türkiye's KVKK), IPD will not be shared. A de-identified minimal dataset supporting the main findings is available as Supplementary File S1; additional de-identified/aggregated data may be provided by the corresponding author upon reasonable request under a data-use agreement.